CLINICAL TRIAL: NCT06865898
Title: Plasma Proteomics Study of End-Stage Liver Disease Patients Based on Olink Technology
Status: Active, not recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202411-016-1
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-09

CONDITIONS: HBV Related Acute-on-chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Exploring Early Biomarkers of Hepatitis B Virus-Related Acute-on-Chronic Liver Failure Using Olink Proteomics

DETAILED DESCRIPTION:
The rationale for this study is that, with the changing epidemiology of liver diseases, traditional diagnostic methods are no longer sufficient to meet clinical needs. Olink technology, however, offers the potential to discover novel biomarkers. By comparing the plasma proteomic profiles of patients with cirrhosis and liver failure, we aim to identify clinically significant markers. This not only has the potential to enhance early diagnostic capabilities but also provides an important basis for personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

* HBV-LC patients were diagnosed based on previous liver biopsy results or clinical evidence and laboratory tests of previous decompensation for more than three months, including ascites, gastrointestinal bleeding, infection, hepatic encephalopathy, or a combination of these symptoms, endoscopic examination (esophageal and gastric varices), and radiological imaging of portal hypertension and/or liver nodules.

The inclusion criteria for HBV-ACHD patients in this study were based on patients with chronic stable decompensated cirrhosis who experienced an acute decompensation within three months. The reference criteria for acute decompensation in the HBV-ACHD group were as follows: patients with previously diagnosed decompensated cirrhosis presenting with a high level of jaundice (total bilirubin ≥5 mg/dL) HBV-ACLF was categorized into three grades based on the severity of the condition. The inclusion criteria for HBV-ACLF-1 were as follows: patients presenting with liver failure alone with an international normalized ratio (INR) ≥1.5 and/or kidney dysfunction and/or hepatic encephalopathy (HE) grade I or II. HBV-ACLF-2 was defined by dual-organ system failure, while HBV-ACLF-3 was characterized by failure involving three or more organ systems.

Exclusion Criteria:

* Associated with other types of hepatitis virus infection or HIV infection, alcoholic liver disease, autoimmune liver disease, drug-induced liver injury; ② Suffering from primary liver cancer or severe heart, digestive, lung, kidney, neurological and psychiatric diseases; ③ Patients with incomplete data and patients unable to participate in the experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with HBV related liver cirrhosis，HBV related acute-on-chronic hepatic dysfunction and HBV related acute-on-chronic liver failure
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days, 90 days

SECONDARY OUTCOMES:
Differential protein levels | 28 days, 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China